CLINICAL TRIAL: NCT05549635
Title: Pulmonary Fibrosis Biobank - Hypersensitivity Pneumonitis
Brief Title: Database and Biobank of Patients With Hypersensitivity Pneumonitis
Acronym: PFBIO-HP
Status: Recruiting | Type: Observational
Sponsor: Nils Hoyer (Other)
Responsible Party: Sponsor-Investigator, Nils Hoyer, Principal Investigator, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Other Study IDs: PFBIO-HP
Record Dates: First submitted 2022-06-13; First posted 2022-09-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Hypersensitivity Pneumonitis
Keywords: biomarker; prognosis; diagnosis; phenotyping; genotyping
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — There will be collected serum, EDTA plasma and DNA from included subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an MDT-diagnosis of hypersensitivity pneumonitis (HP): The overall inclusion criteria of patients in the HP cohort are:
  * Diagnosis of HP at an MDT conference according to the current international guidelines
  * Age of 18 years or older
  * The patients must be capable of giving informed consent

SUMMARY:
Sub-study of the main Pulmonary Fibrosis Biomarker (PFBIO) cohort (NCT02755441), recruiting patients with an MDT-diagnosis of hypersensitivity pneumonitis (HP). Patients are included for the collection of blood samples and regular clinical data.

The database and biobank will be available for studies of HP, and can be directly compared to the main PFBIO cohort, which has recruited patients with Idiopathic pulmonary Fibrosis (IPF) since 2016.

Biomarkers will be assessed as diagnostic and prognostic. Further subtyping of HP, based on blood markers (including precipitins) will also be possible with the PFBIO-HP project.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HP at an MDT conference according to the current international guidelines
* Age of 18 years or older
* The patients must be capable of giving informed consent

Exclusion Criteria:

- Unable to sign informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients with an MDT-diagnosis of HP are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of HP | 0 days
  MDT-Diagnosis of HP
Exposure to inciting antigen (patient reported) | 0 days
  Known exposure, as reported by the patient
Exposure to inciting antigen (measurable) | 0 days
  Measurable exposure, as tested by precipitins
Progression free survival | 3 years
  Survival without progression
Overall survival | 3 years
  Survival after diagnosis

SECONDARY OUTCOMES:
Quality of life questionnaires | 3 years
  SGRQ
Pulmonary function test | 3 years
  FVC
Pulmonary function test | 3 years
  DLCO
Imaging | 3 years
  HRCT scans

CONTACTS AND LOCATIONS:
Locations (1):
- Department of respiratory medicine, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No